CLINICAL TRIAL: NCT01511666
Title: Hyperinvasive Approach to out-of Hospital Cardiac Arrest Using Mechanical Chest Compression Device, Prehospital Intraarrest Cooling, Extracorporeal Life Support and Early Invasive Assessment Compared to Standard of Care. A Randomized Parallel Groups Comparative Study. "Prague OHCA Study"
Brief Title: Hyperinvasive Approach in Cardiac Arrest
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: DSMB recommendation to stop
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Jan Belohlavek, Jan Belohlavek, MD, PhD., Consultant in Cardiology and Critical Care, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prague OHCA study
Record Dates: First submitted 2012-01-13; First posted 2012-01-19 (Estimated); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Out-of Hospital Cardiac Arrest
Keywords: cardiac arrest; mechanical chest compressions; intraarrest cooling; ECLS
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperinvasive arm (Experimental): Hyperinvasive arm encompasses immediate institution of a mechanical chest compression device (LUCAS) and pre-hospital intraarrest cooling by Rhino-Chill device. Immediately after institution of these two devices the patients will be directly transferred to cardiac center cathlab under continuous CPR. The use of drugs and further defibrillations are on a discretion of the emergency physician. After admission to cathlab, overall status, ROSC presence and ECLS inclusion/exclusion criteria will be evaluated.
  Interventions: Device: Prehospital mechanical compressions, intraarrest cooling and in hospital ECLS
- Standard arm (Active Comparator): Patients in standard arm will be further managed as per recent ERC guidelines, ie. continued ACLS. The use of drugs and further defibrillations are on a discretion of the emergency physician. If ROSC is attained, patients will be transferred to the same hospital to one of intensive care units, coronary angiography/PCI will be performed only if indicated according to routine practice and mild therapeutic hypothermia will be instituted as soon as possible as per recent guidelines recommendation.
  Interventions: Other: Standard care

INTERVENTIONS:
Device: Prehospital mechanical compressions, intraarrest cooling and in hospital ECLS — ECLS states for extracorporeal life support.
  Other Names: LUCAS; Rhinochill; ECLS
  Arms: Hyperinvasive arm
Other: Standard care — Standard care as per recent guidelines will be provided.
  Arms: Standard arm

SUMMARY:
Prague out-of Hospital Cardiac Arrest (OHCA) study is a prospective randomized multicenter clinical study comparing use of prehospital intraarrest hypothermia, mechanical chest compression device, extracorporeal life support (ECLS) and early invasive investigation and treatment (coronary angiography/percutaneous coronary intervention [PCI]; pulmonary angiography/percutaneous embolectomy; aortography) in all patients with OHCA of presumed cardiac origin compared to standard of care. It is hypothesized, that above stated "hyperinvasive" approach might improve outcome of out-of hospital cardiac arrest victims.

DETAILED DESCRIPTION:
Background: Out of hospital cardiac arrest (OHCA) has a poor outcome. Recent non-randomized study of ECLS (extracorporeal life support) in OHCA suggested further prospective multicenter studies to define population with OHCA that would benefit from ECLS.

Aim: to perform a prospective randomized multicenter clinical study comparing use of prehospital intraarrest hypothermia, mechanical chest compression device, ECLS and early invasive investigation and treatment (coronary angiography/percutaneous coronary intervention [PCI]; pulmonary angiography/percutaneous embolectomy; aortography) in all patients with OHCA of presumed cardiac origin compared to standard of care.

Planned intervention: patients with witnessed OHCA without ROSC (return of spontaneous circulation) after a minimum of 5 minutes of ACLS by emergency medical service (EMS) team will be after fulfilling of inclusion/exclusion criteria for the study randomized in a 1:1 design to standard vs. hyperinvasive arm. Patients in standard arm will be further managed as per recent guidelines. In hyperinvasive arm, mechanical compression device together with intranasal cooling will be immediately instituted and patients will be transferred to cardiac center directly to cathlab under ongoing CPR. After admission to cathlab, overall status, ROSC and ECLS inclusion/exclusion criteria will be evaluated and in case of no contraindications to ECLS and no ROSC or ROSC with shock, veno-arterial ECLS will be started as soon as possible, not later than 60 minutes after cardiac arrest onset. After ECLS institution, mild hypothermia will be continued by means of ECLS cooling and immediate invasive investigation will be performed in all patients.

Standard postresuscitation care will follow.

ELIGIBILITY:
Inclusion Criteria:

* minimum of 18 and maximum of 65 years
* witnessed out-of-hospital cardiac arrest of presumed cardiac cause
* minimum of 5 minutes of ACLS performed by emergency medical service team without sustained ROSC
* unconsciousness (Glasgow Coma Score < 8)
* ECMO team and bed-capacity in cardiac center available.

Exclusion Criteria:

* OHCA of presumed non-cardiac cause
* unwitnessed collapse
* pregnancy
* sustained ROSC within 5 minutes of ACLS performed by EMS team
* conscious patient
* known bleeding diathesis or suspected or confirmed acute or recent intracranial bleeding
* suspected or confirmed acute stroke
* known severe chronic organ dysfunction or other limitations in therapy
* "do not resuscitate" order or other circumstances making 180 day survival unlikely
* known pre-arrest cerebral performance category CPC ≥ 3.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2020-10-25 (Actual); Study Completion 2020-10-25 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of survival with good neurological outcome (CPC 1-2). | 6 months

SECONDARY OUTCOMES:
Neurological recovery | 30 days
  Neurological recovery will be defined as no or minimal neurological impairment (CPC 1 or 2) at any timepoint within first 30 days after initial cardiac arrest.
Cardiac recovery | 30 days
  Cardiac recovery will be assessed by the clinical status of hemodynamic stability defined as no need for pharmacological or mechanical cardiac support. Systolic function will be measured by echocardiography .

CONTACTS AND LOCATIONS:
Overall Officials: Jan Belohlavek, Principal Investigator — General University Hospital
Locations (1):
- General Teaching Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Smalcova J, Suen J, Huptych M, Franek O, Kavalkova P, Brodska HL, Balik M, Malik J, Pudil J, Smid O, Fajkus M, McInerney MR, Belohlavek J. The significance of possible non-occlusive mesenteric ischemia in relation to neurological outcomes in patients with refractory cardiac arrest - Secondary analysis of the Prague OHCA study. Resuscitation. 2025 Sep;214:110642. doi: 10.1016/j.resuscitation.2025.110642. Epub 2025 May 15. PMID 40381979
- [Derived] Rob D, Farkasovska K, Kreckova M, Smid O, Kavalkova P, Macoun J, Huptych M, Havrankova P, Gallo J, Pudil J, Dusik M, Havranek S, Linhart A, Belohlavek J. Effect of intra-arrest transport, extracorporeal cardiopulmonary resuscitation and immediate invasive assessment in refractory out-of-hospital cardiac arrest: a long-term follow-up of the Prague OHCA trial. Crit Care. 2024 Apr 16;28(1):125. doi: 10.1186/s13054-024-04901-7. PMID 38627823
- [Derived] Smalcova J, Havranek S, Pokorna E, Franek O, Huptych M, Kavalkova P, Pudil J, Rob D, Dusik M, Belohlavek J. Extracorporeal cardiopulmonary resuscitation-based approach to refractory out-of-hospital cardiac arrest: A focus on organ donation, a secondary analysis of a Prague OHCA randomized study. Resuscitation. 2023 Dec;193:109993. doi: 10.1016/j.resuscitation.2023.109993. Epub 2023 Oct 6. PMID 37806620
- [Derived] Dusik M, Rob D, Smalcova J, Havranek S, Karasek J, Smid O, Brodska HL, Kavalkova P, Huptych M, Bakker J, Belohlavek J. Serum lactate in refractory out-of-hospital cardiac arrest: Post-hoc analysis of the Prague OHCA study. Resuscitation. 2023 Nov;192:109935. doi: 10.1016/j.resuscitation.2023.109935. Epub 2023 Aug 11. PMID 37574002
- [Derived] Rob D, Smalcova J, Smid O, Kral A, Kovarnik T, Zemanek D, Kavalkova P, Huptych M, Komarek A, Franek O, Havranek S, Linhart A, Belohlavek J. Extracorporeal versus conventional cardiopulmonary resuscitation for refractory out-of-hospital cardiac arrest: a secondary analysis of the Prague OHCA trial. Crit Care. 2022 Oct 27;26(1):330. doi: 10.1186/s13054-022-04199-3. PMID 36303227
- [Derived] Belohlavek J, Smalcova J, Rob D, Franek O, Smid O, Pokorna M, Horak J, Mrazek V, Kovarnik T, Zemanek D, Kral A, Havranek S, Kavalkova P, Kompelentova L, Tomkova H, Mejstrik A, Valasek J, Peran D, Pekara J, Rulisek J, Balik M, Huptych M, Jarkovsky J, Malik J, Valerianova A, Mlejnsky F, Kolouch P, Havrankova P, Romportl D, Komarek A, Linhart A; Prague OHCA Study Group. Effect of Intra-arrest Transport, Extracorporeal Cardiopulmonary Resuscitation, and Immediate Invasive Assessment and Treatment on Functional Neurologic Outcome in Refractory Out-of-Hospital Cardiac Arrest: A Randomized Clinical Trial. JAMA. 2022 Feb 22;327(8):737-747. doi: 10.1001/jama.2022.1025. PMID 35191923
- [Derived] Belohlavek J, Kucera K, Jarkovsky J, Franek O, Pokorna M, Danda J, Skripsky R, Kandrnal V, Balik M, Kunstyr J, Horak J, Smid O, Valasek J, Mrazek V, Schwarz Z, Linhart A. Hyperinvasive approach to out-of hospital cardiac arrest using mechanical chest compression device, prehospital intraarrest cooling, extracorporeal life support and early invasive assessment compared to standard of care. A randomized parallel groups comparative study proposal. "Prague OHCA study". J Transl Med. 2012 Aug 10;10:163. doi: 10.1186/1479-5876-10-163. PMID 22883307

DOCUMENTS (1):
  • Study Protocol (2012-08-10): https://cdn.clinicaltrials.gov/large-docs/66/NCT01511666/Prot_000.pdf